CLINICAL TRIAL: NCT06088693
Title: The Role of Electroacupuncture With Standard Therapy on Sperm Analysis and SOD Levels in Oligozoospermia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Lisa Yunita, Medical Doctor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 23-06-1010
Record Dates: First submitted 2023-09-11; First posted 2023-10-18 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Oligozoospermia; Oligoasthenozoospermia; Oligoasthenoteratozoospermia
MeSH Terms: conditions — Oligospermia | interventions — Electroacupuncture; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The investigator blind the participant allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients diagnosed with Oligozoospermia who only receive standard therapy from an Andrologist as a standard therapy.
- Intervention (Experimental): Patients diagnosed with Oligozoospermia receive standard therapy from an Andrologist and Electroacupuncture.
  Interventions: Other: Electroacupuncture and Standard Therapy

INTERVENTIONS:
Other: Electroacupuncture and Standard Therapy — Acupuncture Needle Insertion with Electroacupuncture machine.
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to compare in Oligozoospermia Patient. The main questions it aims to answer are: 1. Electroacupuncture therapy and standard therapy can affect oligozoospermia. 2. Electroacupuncture therapy and standard therapy can affect semen and spermatozoa plasma SOD levels.

Researchers will compare patient with standard therapy with patient with standard therapy with electroacupuncture.

DETAILED DESCRIPTION:
1. Male subjects aged more than 25 years and less than 45 years.
2. Oligozoospermia according to the 2010 WHO criteria is mild (10-15 million spermatozoa/mL), moderate (5-10 million spermatozoa/mL) and severe (<5 million spermatozoa/mL).
3. Willing to take part in research and sign informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Male 25 to 45 years old.
* Oligozoospermia according to the 2010 WHO criteria is mild (10-15 million spermatozoa/mL), moderate (5-10 million spermatozoa/mL) and severe (<5 million spermatozoa/mL).
* Willing to participate in research and sign informed consent.

Exclusion Criteria:

* Emergency case patient / bleeding disorders
* Have a tumor, scar tissue or infected wound in the area where the acupuncture needle will be inserted.
* Alcoholic
* Using a pacemaker (heart pacemaker).
* Azoospermia
* Varicocele

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male with Oligozoospermia, Oligoasthenozoospermia, Oligoasthenoteratozoospermia, Oligoteratozoospermia.
Enrollment: 48 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2023-11-26 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Sperm analysis | Before Treatment in day 1, After 30 days of treatment.
  Spermatozoa/mL
SOD Spermatozoa | Before Treatment in day 1, After 30 days of treatment.
  Superokside Dismutase in Spermatozoa
SOD Plasma Semen | Before Treatment in day 1, After 30 days of treatment.
  Superokside Dismutase in Plasma Semen

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Yunita, Principal Investigator — Indonesia University
Locations (1):
- Lisa Yunita, Jakarta, Jakarta Timur, Indonesia

IPD SHARING:
Plan to Share IPD: No